CLINICAL TRIAL: NCT06196060
Title: Improving Theory of Mind in Children With Autism Spectrum Disorder Through Visual Perspective Taking Training: Behavioral and Functional Near-Infrared Spectroscopy Research
Brief Title: Improving ToM in Children With ASD Through VPT Training: Behavioral and fNIRS Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Normal University (Other)
Collaborators: Zhuhai Fudan Innovation Institute (Unknown); Second Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Mi Tian, Associate Professor, Nanjing Normal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNU202202002
Record Dates: First submitted 2023-12-05; First posted 2024-01-09 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Theory of Mind; Visual Perspective Taking; Facial Emotion Recognition
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Visual perspective taking training (Experimental): Participants will receive visual perspective taking training in this arm.
  Interventions: Behavioral: Visual perspective taking training
- Block building training (Experimental): Participants will receive block building training in this arm.
  Interventions: Behavioral: Block building training
- Thought-bubble training (Active Comparator): Participants will receive thought-bubble training in this arm.
  Interventions: Behavioral: Thought-bubble training
- Treatment as usual (Placebo Comparator): Participants will continue to receive routine therapy in this arm.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Visual perspective taking training — Participants will be instructed to utilize small building blocks for the construction of diverse three-dimensional models, with a particular emphasis on employing various perspectives. The visual perspective taking training sessions will be conducted three times weekly over a period of 4 weeks.
  Arms: Visual perspective taking training
Behavioral: Block building training — Participants will be instructed to utilize unit building blocks to construct diverse three-dimensional models. The block building training sessions will be conducted three times weekly over a period of 4 weeks.
  Arms: Block building training
Behavioral: Thought-bubble training — Participants will be instructed in the comprehension of mental states through the utilization of cartoon thought-bubbles as a representational tool. The thought-bubble training sessions will be conducted three times weekly over a period of 4 weeks.
  Arms: Thought-bubble training
Behavioral: Treatment as usual — Participants will continue to receive treatment as usual during the trial.
  Arms: Treatment as usual

SUMMARY:
This study aims to employ a longitudinal tracking research to investigate the effects of a visual perspective taking intervention on the development of theory of mind in children with autism. Additionally, the investigators seek to examine modifications in the neural mechanisms linked to facial emotion recognition in children both before and after intervention by using the functional Near-Infrared Spectroscopy (fNIRS) to record the relative changes in blood oxygen levels in the cerebral cortex with the oddball Face-Periodic Visual Stimulation (FPVS) paradigm.

DETAILED DESCRIPTION:
The deficiency or delayed development of Theory of Mind (ToM) stands as a significant contributing factor to social disorders observed in children with Autism Spectrum Disorder (ASD). Consequently, improving ToM ability is considered pivotal way to improve the development of social function of children with ASD. This study aims to improve ToM ability of children with ASD, and the purpose of this study are as follows:

1. Reveal the development mechanism of theory of mind of children with ASD, based on embodied cognition theory. Explore whether visual perspective taking training can improve the development of Theory of Mind in children with ASD, and if such enhancement exhibits long-term stability.
2. Undertake a longitudinal investigation to assess the stability of visual perspective taking training in improving the development of Theory of Mind in children with ASD. Additionally, the study aims to compare the differential effects and stability of various intervention programs in improving the Theory of Mind in children with ASD.
3. Explore potential disparities in the brain mechanisms of facial emotion recognition between children with ASD and typically developing children before and after the intervention. Specifically, the study seeks to discern whether the intervention can enhance facial emotion recognition abilities in children with ASD and assess the longevity of such enhancements.

The study consists of two parts. In Study 1, participants will be randomly assigned to distinct training groups based on baseline task performance, undergoing three sessions per week for a duration of 4 weeks. In Study 2, the investigators will mainly use the fNIRS with the oddball FPVS paradigm to test children's ability to distinguish facial emotion pictures before and after the intervention, assessing whether the intervention enhances facial emotion recognition ability and if effects vary across different training methods.

ELIGIBILITY:
Inclusion Criteria:

ASD group:

* With a diagnosis of ASD.
* Age between 3 and 8 years old.
* Monolinguals, Chinese native speakers.
* Providing written informed consent sighed by parents.

Control group:

* No diagnosis of ASD (including individuals who are typically developing, have attention deficit hyperactivity disorder, etc.)
* Age between 3 and 8 years old.
* Monolinguals, Chinese native speakers.
* Providing written informed consent sighed by parents.

Exclusion Criteria:

* Language or motor impairments hindering participation in the study.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Theory of Mind scale | The test will be measured before, after immediately and three months after the intervention.
  This scale comprises seven subtests reflecting the sequential development of these concepts throughout the preschool years, including diverse desires, diverse beliefs, knowledge-ignorance or access, contents false belief, explicit false belief, belief emotion and real-apparent emotion.
The Chinese version of Theory of Mind Inventory-2 (ToMI-2-C) | The test will be measured before, after immediately and three months after the intervention.
  The ToMI-2 is a questionnaire filled by parents or guardians. It encompasses 60 items, which are categorized into three empirically derived subscales-Early, Basic, and Advanced-to comprehensively measure ToM abilities.
The Chinese version of Theory of Mind Task Battery (ToMTB) | The test will be measured before, after immediately and three months after the intervention.
  The ToMTB encompasses nine tasks, including an emotion recognition task, a desire-based emotion task, a seeing-leads-to-knowing task and so forth.
Visual perspective taking | The test will be measured before, after immediately and three months after the intervention.
  A small toy will be placed on a square turntable, which has distinct colored sides. The child will be presented with a laminated card representing four images of the toy, each captured from the front, back, left, and right perspectives. The experimenter will randomly place a small doll in different positions (left, right, or the distant side). The child will be asked, 'This is a little seahorse. When the seahorse is here, which view will the seahorse have?' The child's response will be recorded and scored.

SECONDARY OUTCOMES:
Facial emotion recognition | The test will be measured before, after immediately and three months after the intervention.
  fNIRS recordings of relative changes in blood oxygen levels in the cerebral cortex under the oddball FPVS paradigm were employed to assess the recognition of emotional facial images in children with ASD.
Spatial ability | The test will be measured before, after immediately and three months after the intervention.
  Spatial ability will be assessed using the Block Design subtest from the Wechsler Preschool and Primary Scale of Intelligence,4th ed. (WPPSI-IV)
Mental rotation | The test will be measured before, after immediately and three months after the intervention.
  A small toy will be placed on a square turntable, which has distinct colored sides. The child will be presented with a laminated card representing four images of the toy, each captured from the front, back, left, and right perspectives. After the child correctly identifies the starting direction of the toy, the toy will be covered with an opaque cup. Subsequently, the examiner will randomly rotate the turntable by 90 degrees. The child is then tasked with identifying what the toy will look like when the cup is unveiled. The child's response will be recorded and scored.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Zhuhai Fudan Innovation Institute, Zhuhai, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Nanjing Normal University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Caldwell MP, Cheung H, Cheung SK, Li JB, Carrey Siu TS. Visuospatial perspective-taking in social-emotional development: enhancing young children's mind and emotion understanding via block building training. BMC Psychol. 2022 Nov 12;10(1):264. doi: 10.1186/s40359-022-00976-5. PMID 36371295
- [Background] Coll MP, Murphy J, Catmur C, Bird G, Brewer R. The importance of stimulus variability when studying face processing using fast periodic visual stimulation: A novel 'mixed-emotions' paradigm. Cortex. 2019 Aug;117:182-195. doi: 10.1016/j.cortex.2019.03.006. Epub 2019 Mar 19. PMID 30986633
- [Background] Dwyer P, Xu B, Tanaka JW. Investigating the perception of face identity in adults on the autism spectrum using behavioural and electrophysiological measures. Vision Res. 2019 Apr;157:132-141. doi: 10.1016/j.visres.2018.02.013. Epub 2018 Jul 26. PMID 30012353
- [Background] Erle TM, Topolinski S. The grounded nature of psychological perspective-taking. J Pers Soc Psychol. 2017 May;112(5):683-695. doi: 10.1037/pspa0000081. Epub 2017 Mar 2. PMID 28253002
- [Background] Hamilton AF, Brindley R, Frith U. Visual perspective taking impairment in children with autistic spectrum disorder. Cognition. 2009 Oct;113(1):37-44. doi: 10.1016/j.cognition.2009.07.007. Epub 2009 Aug 13. PMID 19682673
- [Background] Hofmann SG, Doan SN, Sprung M, Wilson A, Ebesutani C, Andrews LA, Curtiss J, Harris PL. Training children's theory-of-mind: A meta-analysis of controlled studies. Cognition. 2016 May;150:200-12. doi: 10.1016/j.cognition.2016.01.006. Epub 2016 Feb 20. PMID 26901235
- [Background] Hutchins TL, Prelock PA, Bonazinga L. Psychometric evaluation of the Theory of Mind Inventory (ToMI): a study of typically developing children and children with autism spectrum disorder. J Autism Dev Disord. 2012 Mar;42(3):327-41. doi: 10.1007/s10803-011-1244-7. PMID 21484516
- [Background] Retter TL, Rossion B. Uncovering the neural magnitude and spatio-temporal dynamics of natural image categorization in a fast visual stream. Neuropsychologia. 2016 Oct;91:9-28. doi: 10.1016/j.neuropsychologia.2016.07.028. Epub 2016 Jul 25. PMID 27461075
- [Background] Rossion B. Understanding face perception by means of human electrophysiology. Trends Cogn Sci. 2014 Jun;18(6):310-8. doi: 10.1016/j.tics.2014.02.013. Epub 2014 Apr 1. PMID 24703600
- [Background] Surtees A, Apperly I, Samson D. Similarities and differences in visual and spatial perspective-taking processes. Cognition. 2013 Nov;129(2):426-38. doi: 10.1016/j.cognition.2013.06.008. Epub 2013 Sep 14. PMID 23999408
- [Background] Tian M, Luo T, Ding J, Wang X, Cheung H. Spatial Ability and Theory of Mind: A Mediating Role of Visual Perspective Taking. Child Dev. 2021 Jul;92(4):1590-1604. doi: 10.1111/cdev.13546. Epub 2021 Jan 28. PMID 33507549
- [Background] Tracy JL, Robins RW, Schriber RA, Solomon M. Is emotion recognition impaired in individuals with autism spectrum disorders? J Autism Dev Disord. 2011 Jan;41(1):102-9. doi: 10.1007/s10803-010-1030-y. PMID 20464465
- [Background] Van der Donck S, Dzhelyova M, Vettori S, Mahdi SS, Claes P, Steyaert J, Boets B. Rapid neural categorization of angry and fearful faces is specifically impaired in boys with autism spectrum disorder. J Child Psychol Psychiatry. 2020 Sep;61(9):1019-1029. doi: 10.1111/jcpp.13201. Epub 2020 Jan 31. PMID 32003011
- [Background] Vettori S, Dzhelyova M, Van der Donck S, Jacques C, Steyaert J, Rossion B, Boets B. Reduced neural sensitivity to rapid individual face discrimination in autism spectrum disorder. Neuroimage Clin. 2019;21:101613. doi: 10.1016/j.nicl.2018.101613. Epub 2018 Nov 28. PMID 30522972
- [Background] Wellman HM, Baron-Cohen S, Caswell R, Gomez JC, Swettenham J, Toye E, Lagattuta K. Thought-bubbles help children with autism acquire an alternative to a theory of mind. Autism. 2002 Dec;6(4):343-63. doi: 10.1177/1362361302006004003. PMID 12540127
- [Background] Wellman HM, Liu D. Scaling of theory-of-mind tasks. Child Dev. 2004 Mar-Apr;75(2):523-41. doi: 10.1111/j.1467-8624.2004.00691.x. PMID 15056204
- [Background] Chen KL, Jiang DR, Yu YT, Lee YC. Development and psychometric evidence of the Chinese Version of the Theory of Mind Inventory-2 (ToMI-2) in children with autism spectrum disorder. Research in Autism Spectrum Disorders. 2023; 103: 102132.
- [Background] Kessler K, Wang H. Spatial perspective taking is an embodied process, but not for everyone in the same way: Differences predicted by sex and social skills score. Spatial Cognition & Computation. 2012; 12(2-3): 133-158.
- [Background] Knoll M, Charman T. Teaching false belief and visual perspective taking skills in young children: Can a theory of mind be trained? Child Study Journal. 2000; 30(4): 273-273.
- [Background] Liao Y, Dillenburger K, He W, Xu Y, Cai H. A Systematic Review of Applied Behavior Analytic Interventions for Children with Autism in Mainland China. Review Journal of Autism and Developmental Disorders. 2020; 7(4): 333-351.